CLINICAL TRIAL: NCT07127978
Title: A Prospective, Observational Study Evaluating the Real-World Experience of Givinostat in Patients With Duchenne Muscular Dystrophy
Brief Title: A Study Evaluating the Real-World Experience of Givinostat in Patients With Duchenne Muscular Dystrophy
Acronym: PROVIDUS
Status: Recruiting | Type: Observational
Sponsor: ITF Therapeutics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ITF/2357/62; 126598 (Other: IND Number); 217865 (Other: NDA Number)
Record Dates: First submitted 2025-06-10; First posted 2025-08-17 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Duchene Muscular Dystrophy
Keywords: DMD; DUVYZAT; U.S study; duchenne muscular dystrophy; givinostat; non-interventional study; pediatric neuromuscular disease; rare disease; quality of life; effectiveness; post-marketing requirement; safety; motor function; muscular dystrophy; standard of care; real-world evidence; observational study; post-marketing study
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Rare Diseases; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ambulatory: Ambulatory is defined as being able to complete the 10-meter Walk-Run (10mWR) test within 30 seconds without an assistive device.
  This cohort will include up to 120 patients who are ambulatory prior to starting givinostat treatment.
  Within this cohort , 95 patients must have had prior use or a referral for concomitant use of dystrophin-enhancing therapy (DET), such as exon skipping oligonucleotides or gene therapy.
  Enrollment is capped at 25 patients without prior or referred DET use.
- Non-Ambulatory: Non-ambulatory status is determined by inability to perform the 10mWR test as defined above.
  This cohort will include approximately 180 patients who are non-ambulatory prior to starting givinostat.

SUMMARY:
This is a prospective observational study conducted to evaluate safety, tolerability, and functional outcomes of patients with DMD newly initiating oral givinostat or having started therapy within 6 months as part of routine clinical care in the US. The study has a planned maximum duration of 5 years for the first enrolled patients, including a 24-month enrollment period and a minimum of 2 years of follow-up.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is a rare genetic disorder that leads to progressive muscle degeneration and weakness. Givinostat, an oral histone deacetylase inhibitor, was approved by the FDA in March 2024 for treatment of DMD in patients aged 6 years and older, regardless of mutation type.

Study participation will not influence the course of treatment in any way (including other treatments for DMD), and no treatment will be provided as part of this study. All assessments are intended to be performed at the time of a routine clinical care visit according to clinical practice, and data will be extracted from the medical records.

The FDA is requiring a post-marketing prospective study be conducted for a minimum of 5 years to characterize the incidence, frequency, and severity of thrombocytopenia and serious events of bleeding in patients with DMD treated with oral givinostat in routine clinical practice.

This study is designed as a prospective, observational study to assess safety (including evaluation of AEs of special interest [AESIs]) and effectiveness, in patients with DMD newly initiating oral givinostat as part of routine clinical care in the US in a real-world population. The study will assess AESIs noted above, as well as serious adverse events (SAEs), gastrointestinal (GI) AEs, and dehydration as a sequela to GI AEs. Real-world-treatment patterns of DMD treatments (corticosteroids, exon skipping oligonucleotides and gene therapy) prior to and after givinostat initiation, including treatment duration, and treatment combinations, will be described. Effectiveness evaluations will characterize motor function, quality of life, and activities of daily living in DMD patients treated with givinostat.

The study will enroll 300 participants (180 non-ambulatory and up to 120 ambulatory patients). Participants will be followed for at least two years, with data collected during routine clinical visits. Assessments include lab parameters (e.g., platelet counts, triglycerides), cardiac and pulmonary function, patient-reported outcomes, and motor function scales such as the North Star Ambulatory Assessment (NSAA) and Performance of Upper Limb (PUL) scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any gender at least 6 years of age, diagnosed with DMD (according to genetic test) and have received a prescription for oral givinostat in accordance with the USPI.
* Patient has provided informed consent (and assent when applicable) for participation in the study.
* Patient's index date (first date of givinostat treatment) is no more than 6 months prior to signing of informed consent.
* Patient has the required data available (DMD diagnosis, givinostat administration [dose and schedule], laboratory results [hematology and triglycerides]) for addressing the study objectives for the period between index date and study entry (for patients enrolled after the index date).

Exclusion Criteria:

* Patient previously received givinostat (commercial or investigational product) and permanently discontinued treatment or patient started commercial givinostat for > 6 months before signing of informed consent.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted in the US and plans to enroll 300 patients diagnosed with DMD and treated with givinostat as part of their routine clinical care. Patients will be recruited from expert centers treating DMD patients with specialists in neuromuscular conditions who are routinely involved in the care and treatment of patients with DMD, some of whom would have already gained experience with givinostat.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Characterize the incidence of thrombocytopenia / decreased platelet counts in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Incidence rate of thrombocytopenia (per 100 patient years of observation time) post index date
Characterize the frequency of thrombocytopenia / decreased platelet counts in DMD patients treated with oral givinostat | [Time Frame: From follow up (after first date of givinostat treatment) through end of study (up to 5 years)]
  Frequency and incidence proportion (overall and by maximum severity) of thrombocytopenia
Characterize severity of serious events thrombocytopenia / decreased platelet counts in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Time to first thrombocytopenia event from index date
Characterize the incidence of serious events of bleeding in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Incidence rate of serious bleeding events (per 100-patient years of observation time) post index date
Characterize the frequency of serious events of bleeding in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Frequency and incidence proportion (overall and by maximum severity) of serious bleeding events
Characterize the severity of serious events of bleeding in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Time to first serious bleeding event from index date

SECONDARY OUTCOMES:
Characterize the incidence of other adverse events of special interest (AESIs) in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Incidence rates of each AESI (per 100-patient years of observation time) post index date as well as the incidence proportion of AESIs resulting in dose modifications or givinostat discontinuation
Characterize the frequency other adverse events of special interest (AESIs) in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Frequency and incidence proportion (overall and by maximum severity) of each AESI
Characterize the severity of other adverse events of special interest (AESIs) in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Time to first event of each AESI from index date
Characterize the incidence of all serious adverse events (SAEs) in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Incidence rates of SAEs (per 100-patient years of observation time) post index date by SOC and PT within SOC, and the number of SAEs per patient.
Characterize the frequency of all serious adverse events (SAEs) in DMD patients treated with oral givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Frequency and incidence proportion (overall and by maximum severity) of SAEs (by system organ class [SOC] and preferred term [PT] within SOC), and the frequency and incidence proportion of SAEs resulting in dose modifications or givinostat discontinuation.
Characterize the incidence of gastrointestinal (GI) AEs (nausea, vomiting, diarrhea, abdominal pain, constipation) in DMD patients treated with givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Incidence rates of GI AEs (per 100-patient years of observation time) post index date by PT.
Characterize the frequency of gastrointestinal (GI) AEs (nausea, vomiting, diarrhea, abdominal pain, constipation) in DMD patients treated with givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Frequency and incidence proportion (overall and by severity) of GI AEs (by PT), and frequency and incidence proportion of GI AEs resulting in dose modifications or givinostat discontinuation.
Characterize the severity of gastrointestinal (GI) AEs (nausea, vomiting, diarrhea, abdominal pain, constipation) in DMD patients treated with givinostat | From follow up (after first date of givinostat treatment) through end of study (up to 5 years)
  Number of GI AEs per patient
Characterization of hematology laboratory parameters | From baseline through end of study (up to 5 years)
  Change from baseline hematology laboratory parameters over time
Characterization of triglyceride laboratory parameters | From baseline through end of study (up to 5 years)
  Change from baseline triglyceride laboratory parameters over time

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No